CLINICAL TRIAL: NCT06940622
Title: A Randomized Controlled Trial of D-mannose for the Prophylaxis of Recurrent Urinary Tract Infections in Post-menopausal Women
Brief Title: A Trial of D-mannose for the Prophylaxis of Recurrent Urinary Tract Infections
Acronym: DmannoseRCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Philippe Zimmern, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STU-2024-1090
Record Dates: First submitted 2025-04-11; First posted 2025-04-23 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Recurrent UTIs; Recurrent Urinary Tract Infections; Recurrent Urinary Tract Infections in Women; Recurrent Urinary Tract Infection; Cystitis Recurrent; Cystitis Chronic; UTI; UTI - Urinary Tract Infection; UTI - Lower Urinary Tract Infection
Keywords: D-mannose; dmannose; uti; ruti; recurrent urinary tract infection; urinary tract infection; cystitis; chronic uti; chronic cystitis
MeSH Terms: conditions — Urinary Tract Infections; Cystitis | interventions — Mannose

STUDY DESIGN:
Intervention Model Description: D-mannose and placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- D-mannose (Active Comparator): Dietary Supplement: D-Mannose
  Interventions: Dietary Supplement: D-Mannose
- Placebo (Placebo Comparator): Dietary Supplement: Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: D-Mannose — D-mannose (2g, i.e., 4 x 500mg capsules) daily for 12 months.
  Arms: D-mannose
Dietary Supplement: Placebo — Placebo daily for 12 months.
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, 12-month study to determine the effectiveness of D-mannose (2g daily) supplementation in rUTI (recurrent urinary tract infection) prevention in post-menopausal women.

DETAILED DESCRIPTION:
The proposed study on D-mannose prophylaxis is designed to address a critical unmet medical need to improve the understanding and prevention of rUTI (recurrent urinary tract infection) in post-menopausal women, a population disproportionately affected by rUTI and understudied. The efficacy of D-mannose on preventing uncomplicated rUTI will be elucidated, and additional study measures (including urine culture and one-hour D-mannose test results) may help establish an ideal candidate for responding to daily D-mannose intake over time. The proposed study will follow CONSORT guidelines for randomized clinical trial studies.

Aim 1. Test the hypothesis that D-mannose provides effective rUTI prophylaxis in post-menopausal women over 6 months.

Aim 2. Test the hypothesis that D-mannose provides effective rUTI prophylaxis in post-menopausal women beyond 6 months and up to one year.

The overarching hypotheses are that (1) D-mannose will be found superior to placebo in preventing rUTI in post-menopausal women over 6 months as suggested by one prior RCT7 (Aim 1) and (2) D-mannose will remain effective for rUTI prophylaxis up to one year (Aim 2).

Ninety (90) women currently UTI-free and with a history of uncomplicated rUTI, defined as ≥ 2 symptomatic UTIs in 6 months or ≥ 3 symptomatic UTIs in 12 months, will be enrolled and randomized (2:1 ratio) to receive D-mannose (2g, i.e., 4 x 500mg capsules) or placebo daily for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Female, post-menopausal, age ≥ 55 years old
* Diagnosis of recurrent UTI, defined as ≥ 3 symptomatic culture-proven UTI episodes in 12 months or ≥ 2 in 6 months.
* Currently free from a UTI determined based on absence of symptoms as determined by the UTI symptom assessment questionnaire79 and negative urine culture (<103 colony forming units per ml of urine).
* Able to attend all follow-up appointments for the study.
* A negative upper and lower urinary tract evaluation, including pelvic examination for pelvic organ prolapse (less than stage 2), measurement of post-void residual (less than 50 ml), and imaging (renal ultrasound and standing voiding cystourethrogram) to exclude kidney stone, hydronephrosis, reflux, or urethral diverticulum.

Exclusion Criteria:

* Current use of D-mannose. Patients willing to stop taking D-mannose will be offered to join the trial after a 4-week wash-out period.
* Complicated UTIs, including need for catheter drainage or intermittent catheterization, neurogenic bladder, bladder augmentation, or urinary diversion.
* Ongoing supplement use (Box 1). Patients willing to stop taking the listed supplements will be offered to join the trial after a 4-week wash-out period.
* Evidence of upper tract infection (pyelonephritis), including temperature higher than 38°C, flank/lumbar pain or tenderness
* Diagnosis of interstitial cystitis or overactive bladder syndrome
* Prophylactic antibiotics started in the last 3 months and unwilling to discontinue, or intention to start in the next 12 months
* Use of Uromune or other vaccine approaches to reduce rUTI
* Participation in a research study involving an investigational product in the past 12 weeks
* Receipt of phage treatment
* History of chronic diarrhea requiring regular therapy
* Inability to swallow or known history of gastrointestinal malabsorption
* History of recurrent vaginal yeast infections
* Systemic disease precluding enrollment in this study (uncontrolled diabetes with HgA1C above 7, ongoing chemotherapy or immunotherapy, renal insufficiency [creatinine > 1.5 g/dl]), mental or cognitive impairment, weight loss diet requiring excessively large amounts of fluid intake, or other health-related specific diet).
* Nursing home resident
* BMI >40

Box 1 Supplements to avoid

* Multi-Vitamins and Multi-Mineral capsules
* Specific Vitamins or Minerals (e.g., Calcium, Citrical, Calcium Gummies, Vitamin A, D, Niacin, Pyridoxine, Selenium, Vitamin E, B6, Iron, Omega 3, D3, Magnesium, B-Complex, Women's Ultra MultiVitamin, GNC B-Complex, B-12, PreserVision Areds2, Vitamins D, B Pollen)
* Probiotics
* Cranberry Mannose or Cranberry Extract Weight loss products to avoid
* Medifast
* Vitafusion
* OptiVin Products
* Appetite Suppressants
* Keto-Fuel

Ages: 55 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Failure rate | Through study completion, an average of 5 years
  To determine whether prophylaxis with D-mannose reduces the incidence of UTI episodes compared to placebo. "Failure rate," defined as having 2 UTIs in 6 months or 3 in one year.

SECONDARY OUTCOMES:
Number of UTI antibiotic treatments | Through study completion, an average of 5 years
  To investigate if D-mannose reduces the need for antibiotic use due to recurrent UTIs (measured as number of antibiotic courses for symptomatic culture-proven UTI episodes) compared to placebo.
  Number of UTI antibiotic treatments during the 6 months of treatment. If the participant receives >1 antibiotic course for UTI without symptom relief, it is regarded as one episode and counted as one antibiotic treatment. If there has been an asymptomatic period of at least 14 days in between two UTI antibiotic courses, this will be regarded as a new antibiotic treatment.
Symptom severity | Through study completion, an average of 5 years
  To investigate if D-mannose reduces the severity of UTI symptoms compared to placebo. Record symptom severity using a validated UTI symptom assessment questionnaire.
Serious adverse events associated with D-mannose | Through study completion, an average of 5 years
  To determine the frequency of serious adverse events associated with D-mannose. Number of participants who experienced adverse events >= Grade 3, as defined by Common Terminology Criteria for Adverse Events by CTCA version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Zimmern, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No